CLINICAL TRIAL: NCT02789670
Title: Analysis of the Distribution of Regulatory B Cells in Blood of Multiple Sclerosis Patients
Acronym: B-MS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_35; 2014-A00248-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-05-12; First posted 2016-06-03 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis; Systemic Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to collect peripheral blood mononuclear cells Phenotypic and functional studies using flow cytometric approaches
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MS patients: MS patient group is composed by 20 Individuals with inflammatory brain lesions seen in MRI (Radiologically Isolated syndrome) 20 patients with only one clinically isolated syndrome (CIS) 20 patients with relapsed remittent Multiple sclerosis (RRMS) 20 patients with primary progressive Multiple Sclerosis (PPMS)
  Interventions: Other: Blood sample collection
- Control group patients: Control patient cohort is composed by 20 patients suffering from inflammatory neurological disease other than MS Devic syndrome, Neurosarcoidosis, Neurobehcet... (autoimmune disease control group with neurological disease) 20 patients with systemic sclerosis (autoimmune disease control group) without neurological disease)
  40 healthy subjects
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Peripheral blood will be collected in patients at the different time of the study to analyze phenotypic and functional properties of B cells in MS patients and control group

SUMMARY:
New therapeutic approaches of MS are emerging, targeting different actors of the immune system. Some of them target a specific population of white blood cells: B lymphocytes composed of different subpopulations. The subsets of B cells express different functional properties that control the immune response, but these regulation mechanisms have yet to be clearly described. Some subpopulations could amplify inflammation through IL-6 production for example, whereas some ones contribute to its regulation through the production of IL-10. Using samples collected in a large cohort of individuals with risk of MS and treatment-naive patients in the early onset of the disease, the investigators aim to develop a 2 year follow-up study of the different blood B cells subset distribution and their functional properties in terms of pro- and anti-inflammatory cytokine production in MS. This approach can identify new biomarkers for monitoring of MS patients and lead to better define the indication use of depletive B cell drugs and not to counteract the regulatory action of these cells.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a progressive immuno-inflammatory and degenerative disease of the central nervous system (CNS) and represents the second most common cause of disability in young people. The pathophysiologic mechanisms involved are complex and effective therapeutic strategies have yet to be defined. Moreover it's today evident that treatment approaches have to be performed in a personalized point of view. In this context, biomarkers evaluating the course of the disease but also predicting efficacy of therapy are particularly needed in MS.

Recent data underlines the direct role of B-cells in MS. Such comprehensive data have led to new therapeutic strategies using biotherapies in order to deplete, or modulate, the functions of peripheral B cells. Such approaches have led to contradictory results of efficacy. Today, it remains unclear whether B-cells exert diminished regulatory effects or instead potentiate the pathogenic response of T-cells. Such dual properties may depend on the release of inhibitory (e.g. interleukin-10) or pro-inflammatory cytokines (e.g. interleukin-6) and/or direct interactions with other cells, especially T cells.

The investigators aim to longitudinally evaluate quantitative and functional changes in peripheral blood B-cell subsets (1) at the initiation phases of MS, i.e. radiological isolated syndrome (RIS) and clinically isolated syndrome (CIS) (2) during progression of MS and (3) between the two clinical forms of MS in naïve treatment patient: Relapsing-Remittent MS (RRMS) and Primary Progressive MS (PPMS). B-cell subsets are defined by a combination of membrane markers and enumerated at different time points (inclusion (before treatment) and at 3, 6, 12, 24 months of treatment initiation) in a whole blood flow cytometric (FCM) analysis. The absolute counts and relative proportions of transitional, naïve, memory, and marginal zone-like B-cell subsets are being followed up prospectively in patients with a radiologically isolated syndrome (RIS, n= 20), with clinically isolated syndrome (CIS, n= 20), in MS patients with relapsing remitting form (RRMS, n = 20) and in MS patients with primary progressive evolution of the disease (PPMS, n = 20). Control samples are being collected from patients affected by other inflammatory diseases with neurological symptoms (Devic syndrome, Neurobehcet, neurosarcoidosis n = 20) or without neurological symptoms (systemic sclerosis, SSc, n= 20) and from blood donors (n = 40). In order to evaluate functional properties of B cells, peripheral blood mononuclear cells (PBMC) from each group of patients are activated with CD40 ligand and CpG Oligodeoxynucleotides (CpG ODNs), and IL-10-producing B-cells are enumerated by FCM after a brief incubation with phorbol myristate acetate, ionomycin, and brefeldin A as a protein transport inhibitor agent. In selected CIS and MS patients whose changes in B-cell subpopulations associated with onset or progression of the disease are representative, the B-cell subpopulations will be purified and activated with CD40 ligand and CpG ODNs to be co cultured with anti-CD3-activated autologous T-cells to evaluate inhibitory or potentiating effects on T-cell production of pro-inflammatory cytokines (e.g. IFN-gamma, IL-17).

All phenotypic analyses and cell cultures are performed using previously validated protocols. Our ultimate goal is to correlate quantitative and functional changes of subsets composing the systemic B-cell population with the grading and evolution of MS. Such a strategy could lead to identify which MS patients should receive treatment targeting B cells and when. Further, it may offer a rationale for alternative forms of cell therapy that could introduce for example autologous purified B regulator cells after depletive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS criteria (McDonald et al. 2001) or with Clinically isolated syndrome (CIS) or radiologically isolated syndrome(RIS) or
* Patients patients with other neurological inflammatory disease (OIND) or with autoimmune disease without neurological disease Leroy Metsger' criteria of systemic sclerosis) (OID)

Exclusion Criteria:

* Women without reliable contraception
* Nursing women
* Patients having immunosuppressive treatment in the last month ( beta interféron, glatiramer acetate, natalizumab, fingolimod, glucocorticoid)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the production of IL-10 and IL-6 by B cells in MS patients and the control group at inclusion time point | inclusion
  Percentage of B cells expressing intracellular IL-6 and/or IL-10 will be analyzed in MS patients versus controls at inclusion

SECONDARY OUTCOMES:
Comparison of the production of IL-10 and IL-6 by B cells in MS patients and the control group at the different time points of the study | 3, 6, 12, 24 months
  Percentage of B cells expressing intracellular IL-6 and/or IL-10 will be analyzed in MS patients versus controls at the different time points
Comparison of the production of IL-10 and IL-6 by B cells in the MS patient subgroups at the inclusion time point | inclusion
  Percentage of B cells expressing intracellular IL-6 and/or IL-10 will be analyzed in the different MS patient subgroups at the inclusion time point
Comparison of the production of IL-10 and IL-6 by B cells in the MS patient subgroups at the different time points of the study | 3, 6, 12, 24 months
  Percentage of B cells expressing intracellular IL-6 and/or IL-10 will be analyzed in the different MS patient subgroups at the different time points
Comparison B cell subset distribution in MS patients and the control group | at inclusion
  Distribution of B cell subsets (expressed in percentages) analyzed by flow cytometry in MS and the control group at inclusion time point
Comparison B cell subset distribution | at inclusion
  Distribution of B cell subsets (expressed in absolute values) analyzed by flow cytometry in MS and the control group at inclusion time point
Comparison B cell subset distribution in MS patients versus the control group at the different time points of the study | 3, 6, 12, 24 months
  Distribution of B cell subsets (expressed in percentages) analyzed by flow cytometry in MS and the control group at the different time points of the study
Comparison B cell subset distribution in MS patients versus the control group at the different time points of the study | 3, 6, 12, 24 months
  Distribution of B cell subsets (absolute values) analyzed by flow cytometry in MS and the control group at the different time points of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain DUBUCQUOI, MD PhD, Principal Investigator — CHRU de LILLE
Locations (1):
- CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No